CLINICAL TRIAL: NCT05254652
Title: The Clinical Effect of Pregabalin on Neuropathic Pain in Central Sensitized Patients Who Are Treated With Duloxetine After Total Knee Arthroplasty: Randomized Controlled Trial.
Brief Title: The Clinical Effect of Pregabalin on Neuropathic Pain in Central Sensitized Patients After Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Principal Investigator, Yong In, Professor, The Catholic University of Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KC22MISV0096
Record Dates: First submitted 2022-01-10; First posted 2022-02-24 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Osteoarthritis
Keywords: Pregabalin; neuropathic pain
MeSH Terms: conditions — Osteoarthritis; Neuralgia | interventions — Duloxetine Hydrochloride; Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Duloxetine and Pregabalin (Experimental): Experimental group will take medicine for 10 weeks from 2 weeks before surgery to 8 weeks after surgery. The group takes one pill of duloxetine 30 mg, one pill of pregabalin 150mg after breakfast and one pill of pregabalin 150 mg after dinner.
  Interventions: Drug: Duloxetine 30mg; Drug: Pregabalin 150mg
- Active Comparator: Duloxetine (Active Comparator): Active comparator group will take medicine for 10 weeks from 2 weeks before surgery to 8 weeks after surgery. The group takes only one pill of duloxetine 30 mg after breakfast.
  Interventions: Drug: Duloxetine 30mg

INTERVENTIONS:
Drug: Duloxetine 30mg — Case management consists confirmation of hospital visit date, checking the adverse effect and treatment compliance.
  Other Names: Cymbalta 30mg
Drug: Pregabalin 150mg — Case management consists confirmation of hospital visit date, checking the adverse effect and treatment compliance.
  Other Names: Lyrica 150mg
  Arms: Experimental: Duloxetine and Pregabalin

SUMMARY:
In this study, patients scheduled to undergo total knee arthroplasty (TKA) will be screened through a survey for patients with central sensitivity and patients with neuropathic pain as preoperative evaluation.

It is designed to evaluate the effectiveness of pregabalin with the decision to prescribe duloxetine by dividing patient groups according to central sensitization and neuropathic pain.

DETAILED DESCRIPTION:
Screening for central sensitization and neuropathic pain will be performed two weeks in advance of surgery for patients scheduled to undergo total knee arthroplasty, and is performed through a central sensitization questionnaire and neuropathic pain survey. Through the Central Sensitization Inventory, if the score is 40 or higher out of 100 points, it is considered as the subject of central sensitization. And 13 or higher based on 38 points are considered as the subject of neuropathic pain.

Among the patients who meet these two criteria, only those who agree to the study are targeted. The same probability is assigned by a randomized table two weeks before surgery to a group taking duloxetine and pregabalin and a group taking only duloxetine.

In the case of patients with central sensitization and neuropathic pain, both the experimental group and the control group will take medicine for 10 weeks from 2 weeks before surgery to 8 weeks after surgery. The experimental group takes one pill of duloxetine 30 mg, one pill of pregabalin 150mg after breakfast and one pill of pregabalin 150 mg after dinner. The control group takes only one pill of duloxetine 30 mg after breakfast.

A total of 10 weeks' worth of drugs will be provided two weeks before surgery, and medication compliance will be evaluated based on the number of unused drugs returned by the test subject when the drug is returned. In order to evaluate medication compliance, clinical trials should record the number of drugs provided and returned at each visit and the discontinuation date. Subjects must receive medication guidance on the drug-taking schedule. When the clinical trial is completed or terminated in the middle, the unused or partially used drugs must be returned to the clinical examiner and discarded after confirmation.

Relief drugs can also be taken up to six tablets a day, up to two tablets of 650 mg of Tylenol ER Tablets(acetaminophen) once in both groups.

Anthropological information (gender, age, weight, height, body mass index) and outcome variables (VAS scale for checking the degree of pain) are analyzed for the subjects of the study among patients with central sensitization and neuropathic pain.

The subjects will be collected for three months after surgery in both the experimental group and the control group, and the data will be organized and the results will be derived after the last subject's three-month collection.

From immediately after surgery to three months after surgery, we will evaluate the side effects complaining in the subject group. Side effects will be evaluated through interviews with patients during outpatient visits. The above clinical evaluation is observed during the daily treatment process, and the method performed in this clinical trial is judged to have no unpredictable side effects during the current clinical process.

ELIGIBILITY:
Inclusion Criteria:

* Patients for total knee arthroplasty over the age of 19
* Patients who have the will or ability to follow the doctor's instructions, including rehabilitation treatment such as joint exercise.
* Patients understand this study and agree in writing by the patient's own or by the patient's representative to participate in the study.
* Patients with central sensitization and neuropathic pain.

Exclusion Criteria:

* Rheumatoid arthritis
* Other inflammatory arthritis
* Neuropsychiatric patients
* Hepatic insufficiency
* Renal insufficiency
* Allergy or intolerance to study medications
* Patients with an acetylsalicylic acid of IV (angina, congestive heart failure, dementia, cerebrovascular accident)
* Chronic gabapentin or pregabalin use (regular use for longer than 3 months)
* Chronic opioid use (taking opioids for longer than 3 months)
* Alcohol, drug abuser
* Narcotics addiction

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Visual Pain Scale change | Changes from preoperative Visual pain scale at postoperative 1,2,6,18 weeks and 1 year
  Visual pain scale is a validated questionnaire for evaluation of patients who underwent knee operation. The score range is 0-10. The lower the score, the better the result.

SECONDARY OUTCOMES:
Western Ontario and McMaster University Arthritis Index Scale change | Changes from preoperative Western Ontario and McMaster University Arthritis Index (WOMAC) scale at postoperative 1, 2, 6, 18 weeks and 1 year
  Western Ontario and McMaster University Arthritis Index (WOMAC) scale is a validated questionnarie for evaluation of patients who underwent knee operation. The questionnaire consists of 24 tiems, with five pain-related categories (score range 0-20), two stiffness categories (score range 0-8), and 17 physical functional categories (score range 0-68). All items were scored on a 5-point Likert scale (0 = none, 1 = slightly, 2 = moderate, 3 = serious, 4 = extreme). Total score range is 0-96. The lower the score, the better the result.
Knee range of motion change | Changes from preoperative knee range of motion at postoperative 1, 2, 6, 18 weeks and 1 year
  Knee range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Yong In, MD, PhD, Principal Investigator — The Catholic University of Korea
Locations (1):
- the Catholic Univerisity of Korea Seoul St Mary's hospital, Seoul, South Korea